CLINICAL TRIAL: NCT03325036
Title: Serum Immunological Profiles in Head and Neck Cancer Patients Receiving Curative Radiotherapy: Quantitative Analysis and Prognostic Implication
Brief Title: Serum Immunological Profiles in Head and Neck Cancer Patients Receiving Curative Radiotherapy
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201706046RINC
Record Dates: First submitted 2017-10-24; First posted 2017-10-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2017-07

CONDITIONS: Head and Neck Cancers Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum levels of immunologic profiles — Serum levels of immunologic profiles before and after chemoradiotherapy

SUMMARY:
The purpose of the study is to investigate the clinical usefulness of serum levels of immunologic profiles including pro/anti-inflammatory interleukins, other detectable serum biomarkers including transforming growth factor b1 (TGFb1) or soluble major histocompatibility complex Class I chain-related peptide A (sMICA), and leukocyte subpopulations in head and neck cancers patients receiving curative radiotherapy, as prognostic biomarkers for disease recurrence and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck cancer receiving curative radiotherapy in NTUH radiation therapy department.

Exclusion Criteria:

* Patients with head and neck cancer NOT receiving curative radiotherapy in NTUH radiation therapy department.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Serum levels of immunologic profiles before and after chemoradiotherapy will be prospectively evaluated.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Disease progression | Three years
  Tumor local recurrence or distant metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Ling-Yu Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No